CLINICAL TRIAL: NCT02100228
Title: A Phase Iv Trial To Assess The Effectiveness Of Apixaban Compared With Usual Care Anticoagulation In Subjects With Non-valvular Atrial Fibrillation Undergoing Cardioversion
Brief Title: Study Of The Blood Thinner, Apixaban, For Patients Who Have An Abnormal Heart Rhythm (Atrial Fibrillation) And Expected To Have Treatment To Put Them Back Into A Normal Heart Rhythm (Cardioversion)
Acronym: EMANATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B0661025; CV185-267 (Other: Alias Study Number); 2014-001231-36 (EudraCT Number); EMANATE (Other: Alias Study Number)
Record Dates: First submitted 2014-02-05; First posted 2014-03-31 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
Keywords: apixaban; oral anticoagulant; non-valvular atrial fibrillation; cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental)
  Interventions: Drug: Apixaban
- Parenteral heparin and/or oral Vitamin K antagonist (Active Comparator): Parenteral heparin and/or locally used oral Vitamin K antagonist e.g. warfarin (excludes other novel oral anticoagulants)
  Interventions: Drug: Parenteral heparin and/or oral Vitamin K antagonist

INTERVENTIONS:
Drug: Apixaban — Oral, 2.5 or 5 mg BID
  Arms: Apixaban
Drug: Parenteral heparin and/or oral Vitamin K antagonist — Parenteral heparin and/or locally used oral Vitamin K antagonist e.g. warfarin (excludes other novel oral anticoagulants)
  Arms: Parenteral heparin and/or oral Vitamin K antagonist

SUMMARY:
Some people can develop an abnormal heart beat known as "Atrial fibrillation" or "AF" that puts them at risk of developing clots in the heart. Those clots can travel in the blood circulation to the brain and cause a brain attack ("a stroke"). To prevent those clots forming, blood thinners (anti-coagulants) are used. Apixaban is a blood thinner that works by stopping one of the blood substances required for clotting ("Factor Xa"). It is approved and used to prevent clots forming in people with "AF". Other established blood thinners work by stopping clotting substances being made, known as "Vitamin K antagonists" or "VKAs". An example of this type is Warfarin (Coumadin). The good effects of all blood thinners are preventing clots, and they may also have bad effects of increasing the chance of bleeding. People with "AF", abnormal heart beat, may benefit from changing it back to a normal regular rhythm, known medically as "cardioversion". When this is done, people are currently most commonly treated with a "VKA" blood thinner (e.g. warfarin). The purpose of this study is to assess the good and bad effects ("efficacy" and "safety") of apixaban compared with warfarin in people with "AF" in whom an early cardioversion is planned.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with non-valvular atrial fibrillation (as documented by electrocardiogram (ECG) at Visit 1) indicated for cardioversion and initiation of anticoagulation in accordance with the approved local label. Subjects presenting with atrial flutter with no evidence of atrial fibrillation are not eligible for enrolment.
* Age ≥18 years (Age ≥ 19 years for Korea only and Age ≥ 20 years for Japan only).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or their legally-recognized representative) has been informed of all pertinent aspects of the study.
* The subject is willing to provide contact details for at least one alternate person for study staff to contact regarding their whereabouts, should the subject be lost-to-follow-up over the course of the study. (Subject to IRB/IEC approval)
* Female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28 days after the last dose of assigned treatment. A subject is of childbearing potential if, in the opinion of the investigator, she is biologically capable of having children and is sexually active.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.

Exclusion Criteria:

* Subjects having taken more than 48 hours of an anticoagulant (oral and/or parenteral) immediately prior to randomization.
* Contraindications to apixaban or usual care (eg, VKA) in accordance with the approved local label.
* Severe haemodynamically compromised subjects requiring emergent cardioversion.
* Patients with hemodynamically significant mitral stenosis, mechanical or biological prosthetic valve or valve repair.
* Conditions other than atrial fibrillation that require chronic anticoagulation (eg, a prosthetic heart valve).
* Simultaneous treatment with both aspirin and a thienopyridine (eg, clopidogrel, ticlopidine, prasugrel) or simultaneous treatment with both aspirin and ticagrelor.
* Pregnant females; breastfeeding females; females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after last dose of investigational product.
* Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation. Note: Subjects cannot be randomized into this study more than once.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are BMS/Pfizer employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (165):
- United States (63):
  - Brookwood Medical Center, Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - Integrated Medical Services, Inc./IMS Cardiology, Avondale, Arizona
  - Chula Vista Cardiac Center, Chula Vista, California
  - Hartford Hospital, Hartford, Connecticut
  - Certified Physician Investigator Research Group LLC, Altamonte Springs, Florida
  - Orlando Heart Specialists, Altamonte Springs, Florida
  - The University of Chicago Medical Center Investigational Drug Service Pharmacy (office/storage), Chicago, Illinois
  - The University of Chicago Medical Center Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Franciscan Physician Network-Indiana Heart Physicians, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - UK Good Samaritan Medical Office Building, Lexington, Kentucky
  - Good Samaritan Hospital, Lexington, Kentucky
  - University of Kentucky Medical Center Gill Heart Institute, Lexington, Kentucky
  - University of Kentucky Gill Heart Institute, Lexington, Kentucky
  - University of Kentucky HealthCare/Albert. B, Chandler Hospital, Lexington, Kentucky
  - Aim Clinic, Louisville, Kentucky
  - Cardiology Outpatient Clinic, Louisville, Kentucky
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - University of Massachusetts Worcester Research Pharmacy, Worcester, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hopsital - Allina Health System, Minneapolis, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Missouri Health Care System, Columbia, Missouri
  - University of Missouri Health System, Investigational Drug Serivce, Columbia, Missouri
  - University of Missouri Health System, Columbia, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Electrophysiology Associates, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Robert Wood Johnson Medical School Cardiovascular Institute, New Brunswick, New Jersey
  - State University of New York (SUNY) Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Queens, Flushing, New York
  - Columbia University Medical Center/NY Presbyterian Hospital, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - ProMedica Physicians Cardiology, Oregon, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - ProMedica Physicians Cardiology, Toledo, Ohio
  - Hillcrest Medical Center Pharmacy, Tulsa, Oklahoma
  - Oklahoma Heart Institute at Hillcrest Medical Center, Tulsa, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Cardiology Consultants of Philadelphia, Bristol, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Bryn Mawr Medical Specialist Association, Bryn Mawr, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Cardiology consultants of Philadelphia, Yardley, Pennsylvania
  - Baptist Hospital of Southeast Texas - Beaumont, Beaumont, Texas
  - Southeast Texas Cardiology Associates II, L.L.P., Beaumont, Texas
  - Southeast Texas Cardiology Associates II, L.L.P, Beaumont, Texas
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Utah Cardiology, PC, Layton, Utah
  - Cardiovascular Associates of Virginia-Bon Secours St. Mary's Hospital, Midlothian, Virginia
  - St. Francis Medical Center, Midlothian, Virginia
  - Dominion Cardiovascular Specialists PLLC, Richmond, Virginia
- Belgium (8):
  - Sint-Franciskusziekenhuis, Heusden-Zolder, Limburg
  - University Hospital Ghent, Ghent, Oost-vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Grand Hopital de Charleroi asbl, Gilly
  - Jessa Ziekenhuis-Campus Virga Jesse, Hasselt
  - AZ Delta, Roeselare
  - Cliniques Universitatires UCL Mont-Godinne, Yvoir
- Canada (3):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Institut de Cardiologie de Montreal -ICM / Montreal Heart Institute-MHI, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- Denmark (4):
  - Regionshospitalet Silkeborg, Silkeborg, Central Jutland
  - Slagelse Hospital, Slagelse, Region Sjælland
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Regionhospitalet Viborg, Viborg
- Germany (26):
  - Cardio Centrum Ludwigsburg Bietigheim, Ludwigsburg, Baden-Wurttemberg
  - Charitè Campus Mitte/ Medizinische Klinik mit Schwerpunkt Kardiologie und Angiologie, Berlin
  - Vivantes -Netzwerk fuer Gesundheit GmbH - Klinikum Neukoelln, Berlin
  - Charité - Campus Virchow-Klinikum, Berlin
  - Vivantes Netzwerk fuer Gesundhelt GmbH, Humboldt Klinikum, Berlin
  - Klinikum Links der Weser gGmbH, Bremen
  - Medizinisches Versorgungszentrum am Küchwald GmbH, Chemnitz
  - Klinikum Coburg gGmbH, Coburg
  - Zentrum fuer klinische Pruefungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Praxisklinik Herz und Gefäße, Dresden
  - Johanniter-Krankenhaus Rheinhausen GmbH/ Klinik fuer Kardiologie, Duisburg
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Johann-Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Universitatsmedizin Greifswald, Greifswald
  - Universitätsklinikum Hamburg Eppendorf, Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Unklinik Heidelberg, Heidelberg
  - Klinikum Heidenheim, Heidenheim
  - Klinikum Ingolstadt/ Medizinische Klinik I und IV, Ingolstadt
  - Cardiocenter Rhythmologie, Leipzig
  - Herzzentrum Leipzig GmbH/ Abteilung für Rhythmologie, Leipzig
  - Katholisches Klinikum Mainz, Mainz
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Universitaetsklinikum Tuebingen, Tübingen
  - Prof. Dr. med. Werner Jung,Schwarzwald - Baar Klinikum, Villingen-Schwenningen
  - Josephs-Hospital Warendorf, Warendorf
- Israel (15):
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center (Cardiology), Ashkelon
  - Soroka University Medical Centre, Soroka Medical center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Mount Scopus, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - ZIV Medical Center, Safed
  - Clinical Trial Network Services, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Baruch Padeh Medical Center, Tiberias
- Italy (8):
  - Ospedale Generale Regionale F. Miulli-Ente Ecclesiastico, Acquaviva Delle Fonti (BA), BARI
  - Policlinico Universitario Campus Biomedico, Rome, Lazio
  - I.R.C.C.S. Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Torrette Di Ancona, The Marches
  - Presidio Ospedaliero San Donato, Arezzo
  - Azienda Ospedaliero Universitaria Careggi, Medicina e Cardiologia Geriatrica, Florence
  - Centro Cardiologico Monzino, Milan
  - DAI Malattie Cardiovascolari e Respiratorie, Roma
- Japan (4):
  - Tosei General Hospital, Seto, Aichi-ken
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Osaka General Medical Center, Osaka
  - Nippon Medical School Hospital, Tokyo
- Romania (8):
  - Brasov Emergency Clinical County Hospital, Brasov
  - "Prof. Dr.C.C. lliescu" Emergency Institute for Cardiovascular Diseases Bucharest, Bucharest
  - Bucharest Emergency University Hospital, Bucharest
  - Cluj-Napoca Rehabilitation Clinical Hospital, Cluj-Napoca
  - Craiova Emergency Clinical County Hospital, Craiova
  - Prof.Dr.George I.M. Georgescu Cardiovascular Diseases Institute, Iași
  - Cardio Med SRL, Târgu Mureş
  - Tirgu Mures Emergency Clinical County Hospital, Târgu Mureş
- South Korea (12):
  - Korea University Guro Hospital, Seoul, Korea, Republic of
  - Dong-A Unversity Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Hospital, Deagu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, cardiology and Electrophysiology, Seoul
  - The Catholic University of Korea Seoul ST.MARY'S Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Division of Cardiology, Suwon
- Spain (7):
  - Hospital Universitario San Juan de Alicante, San Juan, Alicante
  - Hospital de Sierrallana, Torrelavega, Cantabria
  - Consorci Sanitari de Terrassa Hospital de Terrassa, Terrassa, Catalonia
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital de Basurto, Bilbao
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Fundacion Jimenez Diaz, Madrid
- Sweden (7):
  - Danderyds Sjukhus AB, Stockholm, Södermanland County
  - Akademiska Sjukhuset I Uppsala/ Kardiologikliniken, Uppsala, Uppsala IAN
  - Sahlgrenska University Hospital, Gothenburg
  - Linkopings Universitetssjukhus Kardiologkliniken, Linköping
  - Universitetssjukhuset i Orebro/ Hjartmottagningen, Örebro
  - Skelleftea Country Hospital, Skellefteå
  - Sodersjukhuset, Stockholm

REFERENCES:
- [Derived] Ezekowitz MD, Pollack CV Jr, Halperin JL, England RD, VanPelt Nguyen S, Spahr J, Sudworth M, Cater NB, Breazna A, Oldgren J, Kirchhof P. Apixaban compared to heparin/vitamin K antagonist in patients with atrial fibrillation scheduled for cardioversion: the EMANATE trial. Eur Heart J. 2018 Aug 21;39(32):2959-2971. doi: 10.1093/eurheartj/ehy148. PMID 29659797
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661025&StudyName=A%20Phase%20IV%20Trial%20To%20Assess%20The%20Effectiveness%20Of%20Apixaban%20Compared%20With%20Usual%20Care%20Anticoagulation%20In%20Subjects%20With%20Non-Valvular%20Atrial%20Fibrillation%20Undergoing%20Cardioversion

RESULTS

PARTICIPANT FLOW:
Groups:
- Apixaban: Participants with non-valvular atrial fibrillation undergoing cardioversion, received Apixaban orally for 30 days after cardioversion or 90 days after randomization if cardioversion was not performed. The dosing of Apixaban was based on investigator's judgement as per local label for the prevention of stroke and systemic embolism in participants.
- Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care): Participants with non-valvular atrial fibrillation undergoing cardioversion, received parenteral heparin and/or oral Vitamin K antagonist as usual care, orally for 30 days after cardioversion or 90 days after randomization if cardioversion was not performed. The dosing of the parenteral heparin and Vitamin K antagonist was based on individual participant's sensitivity to the drug according to the investigators usual practice.
Period: Overall Study
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Started | 753 (735 treated with Apixaban) | 747 (721 treated with Usual Care)
Completed | 678 | 657
Not Completed | 75 | 90
Not completed — Other | 19 | 19
Not completed — Administrative reason | 0 | 1
Not completed — Inclusion/Exclusion criteria not met | 12 | 16
Not completed — Non-compliance | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 27 | 37
Not completed — Adverse Event | 16 | 12
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care) | Total
Number analyzed (Participants) | 753 | 747 | 1500
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.19) | 64.5 (12.76) | 64.6 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 250 | 498
  Male | 505 | 497 | 1002
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 100 | 99 | 199
  Unknown or Not Reported | 645 | 639 | 1284
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 654 | 648 | 1302
  Black or African American | 21 | 20 | 41
  Asian | 78 | 76 | 154
  Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Stroke Event
Description: An acute stroke was defined as a new, important neurological insufficiency of rapid onset that lasted for at least 24 hours and that was not due to a readily identifiable non-vascular cause (like brain tumor or trauma).
Time Frame: Baseline up to 30 days post cardioversion (or up to 90 days after randomization, if cardioversion was not performed within that time frame)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 753 | 747
participants | 0 | 6
Statistical Analysis 1: Comparison: Apixaban vs Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care); Display exact confidence limits for relative risk and Fisher's exact test for comparisons of two proportions; Test type: Superiority — This was a descriptive study, and there was no formal pre-defined hypothesis testing; p = 0.0151, Fisher Exact — nominal p-value; Risk Ratio (RR) = 0.0000, 95% CI 2-sided [0.0000 to 0.6425]

2. Primary Outcome: Number of Participants With Systemic Embolism Event
Description: Systemic embolism occurred in participant when there was a clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries), which was supported by evidence of embolism from surgical specimens, autopsy, angiography, or other objective testing.
Time Frame: as for outcome 1
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 753 | 747
participants | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Number of Participants With Major Bleeding Event
Description: Major bleeding was defined as clinically evident bleeding that was accompanied by one or more of the following: a decrease in hemoglobin of 2 gram per deciliter or more, a transfusion of 2 or more units of packed red blood cells, bleeding that was fatal or bleeding that occurred in at least one of the following critical sites: intracranial, intra-spinal, intraocular (within the corpus of the eye; thus, a conjunctival bleed was not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal.
Time Frame: as for outcome 1
Population: Safety data set included all treated participants (randomized participants who received at least one dose of study drug).
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 735 | 721
participants | 3 | 6
Statistical Analysis 1: Comparison: Apixaban vs Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care); Display exact confidence limits for relative risk and Fisher's exact test for comparisons of two proportions; Test type: Superiority — This was a descriptive study, and there was no formal pre-defined hypothesis testing; p = 0.3378, Fisher Exact — nominal p-value; Risk Ratio (RR) = 0.4905, 95% CI 2-sided [0.1046 to 2.0678]

4. Primary Outcome: Number of Participants With Clinically Relevant Non-Major Bleeding Events
Description: Clinically relevant non-major bleeding was defined as the clinically evident bleeding that consisted of any bleeding that compromised hemodynamics, that led to hospitalization, subcutaneous hematoma larger than 25/100 centimeter square if there was a traumatic cause, intramuscular hematoma documented by ultrasonography, epistaxis, gingival bleeding occurred spontaneously, hematuria that was macroscopic and was spontaneous, macroscopic gastrointestinal hemorrhage included at least one episode of melena or hematemesis, rectal blood loss, hemoptysis or any other bleeding type considered to have clinical consequences for a participant, such as medical intervention, the need for unscheduled contact with a physician, or temporary cessation of a study drug, or associated with pain or impairment of activities of daily life.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 735 | 721
participants | 11 | 13
Statistical Analysis 1: Comparison: Apixaban vs Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care); Display exact confidence limits for relative risk and Fisher's exact test for comparisons of two proportions; Test type: Superiority — This was a descriptive study, and there was no formal pre-defined hypothesis testing; p = 0.6851, Fisher Exact — nominal p-value; Risk Ratio (RR) = 0.8300, 95% CI 2-sided [0.3433 to 1.8916]

5. Primary Outcome: Number of Participants With All Cause Death
Time Frame: as for outcome 1
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 753 | 747
participants | 2 | 1
Statistical Analysis 1: Comparison: Apixaban vs Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care); Display exact confidence limits for relative risk and Fisher's exact test for comparisons of two proportions; Test type: Superiority — This was a descriptive study, and there was no formal pre-defined hypothesis testing; p > 0.9999, Fisher Exact — nominal p-value; Risk Ratio (RR) = 1.9841, 95% CI 2-sided [0.1866 to 53.9968]

6. Secondary Outcome: Time to First Attempt of Cardioversion
Description: Cardioversion was an effective method of converting an abnormally fast heart rate (tachycardia) or other cardiac arrhythmia to normal rhythm using electricity or drugs. First attempt of cardioversion was defined as the first time the participant was admitted for the cardioversion procedure.
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: Full analysis set included all randomized participants. Here, "N" (number of participants analyzed) signifies participants who were evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 510 | 511
days | 2.0 [1 to 93] | 2.0 [1 to 126]

7. Secondary Outcome: Number of Participants With Different Type of Cardioversion Events
Description: Cardioversion was an effective method of converting an abnormally fast heart rate (tachycardia) or other cardiac arrhythmia to normal rhythm using different type of cardioversion events i.e. electrical and pharmacologic. Electrical cardioversion was a procedure in which an electric current was used to reset the heart's rhythm back to its regular pattern (normal sinus rhythm). Pharmacologic cardioversion, also called chemical cardioversion, used antiarrhythmia medication instead of an electrical shock.
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: Full analysis set included all randomized participants. Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 496 | 494
participants
  Electrical | 461 | 464
  Pharmacologic | 35 | 30

8. Secondary Outcome: Number of Cardioversion Attempt of Participants
Description: Cardioversion attempts were defined as the number of times the participant was admitted to hospital for the cardioversion procedure and not the number of attempts during a single hospital admission.
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 753 | 747
participants
  No Cardioversion Attempt | 234 | 224
  1 Cardioversion Attempt | 488 | 496
  More than 2 Cardioversion Attempts | 31 | 27

9. Secondary Outcome: Number of Participants With Their Rhythm Status
Description: Rhythm status was further distinguished into sinus rhythm, atrial fibrillation and atrial flutter. Sinus rhythm was defined as a normal heartbeat. Atrial fibrillation was an irregular heartbeat (arrhythmia) that can lead to blood clots, stroke, heart failure and other heart-related complications and atrial flutter was a common abnormal heart rhythm that was usually associated with a fast heart rate (100 or more heart beats per minute).
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: Safety data set included all treated participants (randomized participants who received at least one dose of study drug). Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 719 | 712
participants
  Normal Sinus | 1 | 2
  Atrial Fibrillation | 715 | 704
  Atrial Flutter | 3 | 6

10. Secondary Outcome: Duration of Hospital Stay of Participants
Description: Duration of hospital stay was defined as the number of hours from hospital admission to hospital discharge followed by early cardioversion.
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 330 | 346
hours | 45.36 [0.4 to 747.0] | 49.47 [0.6 to 709.6]

11. Secondary Outcome: Number of Participants Who Used Image Guidance Approach
Description: An image-guided approach helped cardioversion earlier than the conventional minimum of 3 weeks of anticoagulation that would normally be required prior to cardioversion. Transesophageal echocardiography (TEE or TOE) and computed tomography (CT) were 2 image-guided approaches that were used in this study.
Time Frame: Baseline up to Day of first attempt of cardioversion procedure (Visit 2, up to 130 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
Number analyzed (Participants) | 753 | 747
participants | 383 | 399

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after cardioversion or 90 days after randomization, if cardioversion was not performed
Description: Same event may appear as adverse event (AE) and serious adverse event (SAE), what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety data set included all treated participants.
Arm/Group | Apixaban | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care)
All-Cause Mortality (participants affected / at risk) | 1/735 | 3/721
Serious Adverse Events (participants affected / at risk) | 100/735 | 112/721
Other Adverse Events (participants affected / at risk) | 70/735 | 101/721
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=735) | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care) (N=721)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 2 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 27 | 40
ATRIAL FLUTTER (Cardiac disorders) | 3 | 6
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 3
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR DISSOCIATION (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 5 | 7
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 9 | 7
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 2 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 6
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
MITRAL VALVE PROLAPSE (Cardiac disorders) | 0 | 3
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
PERICARDITIS CONSTRICTIVE (Cardiac disorders) | 1 | 0
SINUS ARREST (Cardiac disorders) | 2 | 1
SINUS NODE DYSFUNCTION (Cardiac disorders) | 2 | 1
TACHYARRHYTHMIA (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0
TACHYCARDIA INDUCED CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
ADENOMATOUS POLYPOSIS COLI (Congenital, familial and genetic disorders) | 1 | 0
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1 | 1
ADRENAL HAEMORRHAGE (Endocrine disorders) | 1 | 0
TOXIC NODULAR GOITRE (Endocrine disorders) | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 1
FEMORAL HERNIA INCARCERATED (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 0 | 1
MESENTERIC PANNICULITIS (Gastrointestinal disorders) | 1 | 0
OEDEMATOUS PANCREATITIS (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
HERNIA (General disorders) | 1 | 0
MUCOSAL HAEMORRHAGE (General disorders) | 0 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 0
SUDDEN DEATH (General disorders) | 0 | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 0
HEPATIC CONGESTION (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0
CELLULITIS (Infections and infestations) | 1 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
INTESTINAL SEPSIS (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 5
SEPSIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
UROSEPSIS (Infections and infestations) | 0 | 1
ARTERIAL BYPASS THROMBOSIS (Injury, poisoning and procedural complications) | 0 | 1
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 3
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 1
COMPUTERISED TOMOGRAM CORONARY ARTERY ABNORMAL (Investigations) | 1 | 0
FUNCTIONAL RESIDUAL CAPACITY DECREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN INJURY (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 3
DEMENTIA (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 2
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 2
DEPRESSION (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 5
HAEMATURIA (Renal and urinary disorders) | 0 | 1
POSTRENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
MEDIASTINAL CYST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY SARCOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 2
HYPOTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=735) | Parenteral Heparin/Oral Vitamin K Antagonist (Usual Care) (N=721)
ATRIAL FIBRILLATION (Cardiac disorders) | 43 | 46
ATRIAL THROMBOSIS (Cardiac disorders) | 17 | 13
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 0 | 19
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 27
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 | 8

LIMITATIONS AND CAVEATS:
The prioritization of outcome measures is not mentioned in the study documents (Statistical Analysis Plan and Protocol). The prioritization of outcome measures is based on team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT02100228/SAP_000.pdf
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT02100228/Prot_001.pdf